CLINICAL TRIAL: NCT00842673
Title: A Double-Blind Placebo-Controlled Preliminary Study of the Efficacy, Safety and Tolerability of ST101 Tablets in the Treatment of Alzheimer's Disease
Brief Title: Preliminary Efficacy and Safety Study of ST101 in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sonexa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST101-A001-201
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Alzheimer Type Senile Dementia; Cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 30 mg ST101
  Interventions: Drug: ST101
- 2 (Experimental): 90 mg ST101
  Interventions: Drug: ST101
- 3 (Experimental): 180 mg ST101
  Interventions: Drug: ST101
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ST101 — 30 mg; administered once/day
  Arms: 1
Drug: ST101 — 90 mg; administered once/day
  Arms: 2
Drug: ST101 — 180 mg; administered once/day
  Arms: 3
Drug: Placebo — placebo to match ST101 tablets
  Arms: 4

SUMMARY:
This study will investigate the ability of ST101 to improve memory in people with Alzheimer's disease. This study also will examine the safety and tolerability of the drug. This study is evaluating 3 different dose levels of ST101 and placebo. Patients will have a 1 in 4 chance of getting placebo.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive and fatal neurological illness. It produces changes in the brain that include loss of cells and accumulation of abnormal protein deposits. Initial symptoms are cognitive, with deficiencies in short-term memory the most common symptom. As the disease progresses so does the severity of cognitive deficiency. Loss of speech and immobility occur in the terminal stages There is no cure for AD and no marketed treatment that modifies the underlying disease process. Available therapies improve some symptoms of AD by increasing brain concentrations of molecules involved in cognition. ST101 differs from marketed therapies in that it has demonstrated two actions in animal research testing. It improves cognition and it also reduces the accumulation of abnormal protein deposits in the brain. These two properties suggest that ST101 may be a promising agent for the treatment of AD. This study is designed as a preliminary dose exploration/proof-of-concept investigation of the ability of ST101 to improve cognition during 12 weeks of administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic evidence of mild to moderate Alzheimer's disease.
* CT or MRI results within the past 12 months that rule out dementia due to non-Alzheimer's etiology.
* A reliable and capable caregiver.

Exclusion Criteria:

* Subjects who reside in a skilled nursing facility.
* Subjects with B12 or folate deficiency.
* Subjects with chronic hepatic disease.
* Subjects with a recent history of hematologic/oncologic disorders.
* Subjects who have experienced a myocardial infarction with the past year.
* Dementia caused or complicated by other organic disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-cog) | Baseline, 4 weeks, 8 weeks,12 weeks

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | Baseline, 4 weeks, 8 weeks, 12 weeks
Neuropsychiatric Inventory (NPI) | Baseline, 4 weeks, 8 weeks, 12 weeks
Alzheimer's Disease Cooperative Study- Clinical Global Impression (ADCS-CGI) | Baseline (severity); 4 weeks, 8 weeks, 12 weeks (change)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (15):
  - Costa Mesa, California
  - Redlands, California
  - San Diego, California
  - Walnut Creek, California
  - Deerfield Beach, Florida
  - Delray Beach, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Durham, North Carolina
  - Toledo, Ohio
  - Jenkinton, Pennsylvania
  - Wichita Falls, Texas
  - Bennington, Vermont
- Canada (3):
  - Peterborough, Ontario
  - Toronto, Ontario
  - Montreal, Quebec